CLINICAL TRIAL: NCT00606385
Title: Prospective Randomized Trial of Laparoscopic Versus Open Liver Resection for Patients With Hepatocellular Carcinoma
Brief Title: Prospective Randomized Trial of Laparoscopic Versus Open Liver Resection for HCC
Acronym: HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho-Seong Han, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-GS-HBP1; SNUBH-GS-HBP1 (Other: Ministry Of Food And Drug Safety)
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Recurrence; Survival; Immunology; Laparoscopy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic liver resection (Experimental): Patients who underwent laparoscopic liver resection for HCC
  Interventions: Procedure: Liver resection
- open liver resection (Active Comparator): Patients who underwent open liver resection for HCC
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Laparoscopic or Open hepatectomy

SUMMARY:
Short-term outcomes of laparoscopic liver resection is better than those of open liver resection

Laparoscopic liver resection is better than open resection in immunological aspects

DETAILED DESCRIPTION:
Advantages and disadvantages of the laparoscopic compared with the open approach for liver resections

1. Advantages 1) Less postoperative ascites production 2) Reduced postoperative pain 3) Feasible in selected cirrhotics who have contraindications to open surgery 4) Less intra-abdominal adhesions (easier salvage transplantation) 5) Shorter recovery time 6) Shorter length of stay 7) Reduced financial cost
2. Disadvantages 1) No manual palpation or exploration of the liver parenchyma possible (with the pure laparoscopic approach) 2) High demand in surgical skill (especially major resections)

ELIGIBILITY:
Inclusion Criteria:

* Radiologically diagnosed hepatocellular carcinoma
* Child classification A or B
* Aged 20 to 80
* Informed consent taken

Exclusion Criteria:

* Child classification C
* Extrahepatic metastasis
* Tumor located in central area or adjacent to middle hepatic vein
* Recurred hepatocellular carcinoma
* Critically ill patient
* Patient with psychiatric disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years after operation

SECONDARY OUTCOMES:
Survival | 2 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Han, MD, PhD, Study Chair — Department of Surgery, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon YS, Han HS, Choi YS, Jang JY, Suh KS, Kim SW, Lee KU, Park YH. Total laparoscopic right posterior sectionectomy for hepatocellular carcinoma. J Laparoendosc Adv Surg Tech A. 2006 Jun;16(3):274-7. doi: 10.1089/lap.2006.16.274. PMID 16796440
- [Background] Min SK, Han HS, Kim SW, Park YH, Lee HO, Lee JH. Initial experiences with laparoscopy-assisted and total laparoscopy for anatomical liver resection: a preliminary study. J Korean Med Sci. 2006 Feb;21(1):69-74. doi: 10.3346/jkms.2006.21.1.69. PMID 16479068
- [Background] Yoon YS, Han HS, Choi YS, Lee SI, Jang JY, Suh KS, Kim SW, Lee KU, Park YH. Total laparoscopic left lateral sectionectomy performed in a child with benign liver mass. J Pediatr Surg. 2006 Jan;41(1):e25-8. doi: 10.1016/j.jpedsurg.2005.10.068. PMID 16410084